CLINICAL TRIAL: NCT04994067
Title: Intra-Operative Radiation Therapy (IORT) Using the IntraBeam® System - A Registry Protocol
Brief Title: Intra-Operative Radiation Registry
Status: Recruiting | Type: Observational
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-9409
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: intraoperative radiation therapy; partial breast irradiation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This registry trial is designed to track the local control rates and side effects of IORT, which will be implemented for women who are suitable partial breast irradiation (PBI) per the latest American Society of Radiation Oncology (ASTRO) guidelines.

DETAILED DESCRIPTION:
Eligible patients will be referred for radiation oncology consultation by the operating surgeon. Patients will be presented with all radiation options and if they choose IORT, they will be offered enrollment onto the registry trial and consented accordingly. The registry will collect treatment data from the operation, radiation and pathology notes post IORT for each patient enrolled. Sources of research material, i.e. resected breast tissue and lymph nodes, will be obtained as part of routine clinical care. No additional tissue will be collected from patients due to enrollment on this registry trial. No additional studies will be performed outside of the routine standard of care.

Post treatment, the registry will collect data based on the standard of care follow up schedule. Follow-up visits will be scheduled 2-3 weeks post-operatively, as per standard of care, to review the final pathology and for the initial toxicity assessment. Patients found to have positive margins and/or lymph node involvement may require further surgery and/or additional external beam radiation. Additional follow-up visits with radiation oncology will be scheduled at 6 months and 1, 2, 3, 4, and 5 years following IORT. Toxicity will be scored using Common Terminology Criteria for Adverse Events (CTCAE) v4.03. Local control will be evaluated using clinical exam and semi-annual to annual mammograms. All such information will be tracked and recorded into the registry database.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Age ≥ 45
* cT1-2N0, <3.5cm invasive breast cancer, estrogen-receptor positive or DCIS of breast, Grade 1-2, mammographically detected, < 2.5 cm, estrogen-receptor positive
* Suitable for breast conserving surgery
* No contraindication to radiation
* Mammogram within 6 months of planned procedure
* Fitness for lumpectomy under general anesthesia
* Planned to receive IORT

Exclusion criteria

* Known axillary lymph node positive breast cancer (negative biopsy not required)
* Multicentric cancer in the same breast as diagnosed by clinical examination, mammography, ultrasound, MRI or pathologic assessment, not amenable to excision with negative margins with a single lumpectomy.
* Patients known to have BRCA 1/2 (breast cancer 1, breast cancer 2) gene
* Patients undergoing neoadjuvant chemotherapy
* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Patients enrolled on this study will be planned for lumpectomy with or without sentinel node biopsy for early stage breast cancer. Patients will be evaluated by a radiation oncologist who specializes in the treatment of breast cancer and will be deemed to be eligible for IORT. Patients with a history of ipsilateral cancer and/or prior in-field radiation are eligible, as IORT would likely be less toxic than repeat whole or partial breast external beam radiation and can allow patients to avoid mastectomy who wish to do so.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-08-09 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2032-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients with locally controlled disease | 5 years following radiation therapy
  How many patients have recurrent disease following intra-operative radiation
Number of patients with regionally controlled disease | 5 years following radiation therapy
  How many patients have recurrent nodal disease following intra-operative radiation
Number of patients with grade 2 or higher toxicities | 5 years following radiation therapy
  How many patients have toxicity as measured by the CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Jana Fox, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center - Moses Campus, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clarke M, Collins R, Darby S, Davies C, Elphinstone P, Evans V, Godwin J, Gray R, Hicks C, James S, MacKinnon E, McGale P, McHugh T, Peto R, Taylor C, Wang Y; Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Effects of radiotherapy and of differences in the extent of surgery for early breast cancer on local recurrence and 15-year survival: an overview of the randomised trials. Lancet. 2005 Dec 17;366(9503):2087-106. doi: 10.1016/S0140-6736(05)67887-7. PMID 16360786
- [Background] Smith TE, Lee D, Turner BC, Carter D, Haffty BG. True recurrence vs. new primary ipsilateral breast tumor relapse: an analysis of clinical and pathologic differences and their implications in natural history, prognoses, and therapeutic management. Int J Radiat Oncol Biol Phys. 2000 Dec 1;48(5):1281-9. doi: 10.1016/s0360-3016(00)01378-x. PMID 11121624
- [Background] Polgar C, Fodor J, Major T, Nemeth G, Lovey K, Orosz Z, Sulyok Z, Takacsi-Nagy Z, Kasler M. Breast-conserving treatment with partial or whole breast irradiation for low-risk invasive breast carcinoma--5-year results of a randomized trial. Int J Radiat Oncol Biol Phys. 2007 Nov 1;69(3):694-702. doi: 10.1016/j.ijrobp.2007.04.022. Epub 2007 May 25. PMID 17531400
- [Background] King TA, Bolton JS, Kuske RR, Fuhrman GM, Scroggins TG, Jiang XZ. Long-term results of wide-field brachytherapy as the sole method of radiation therapy after segmental mastectomy for T(is,1,2) breast cancer. Am J Surg. 2000 Oct;180(4):299-304. doi: 10.1016/s0002-9610(00)00454-2. PMID 11113440
- [Background] Vicini FA, Baglan KL, Kestin LL, Mitchell C, Chen PY, Frazier RC, Edmundson G, Goldstein NS, Benitez P, Huang RR, Martinez A. Accelerated treatment of breast cancer. J Clin Oncol. 2001 Apr 1;19(7):1993-2001. doi: 10.1200/JCO.2001.19.7.1993. PMID 11283132
- [Background] Kaufman SA, DiPetrillo TA, Price LL, Midle JB, Wazer DE. Long-term outcome and toxicity in a Phase I/II trial using high-dose-rate multicatheter interstitial brachytherapy for T1/T2 breast cancer. Brachytherapy. 2007 Oct-Dec;6(4):286-92. doi: 10.1016/j.brachy.2007.09.001. PMID 17991625
- [Background] Arthur DW, Winter K, Kuske RR, Bolton J, Rabinovitch R, White J, Hanson WF, Wilenzick RM, McCormick B. A Phase II trial of brachytherapy alone after lumpectomy for select breast cancer: tumor control and survival outcomes of RTOG 95-17. Int J Radiat Oncol Biol Phys. 2008 Oct 1;72(2):467-73. doi: 10.1016/j.ijrobp.2007.12.056. Epub 2008 Mar 4. PMID 18294778
- [Background] Rabinovitch R, Winter K, Kuske R, Bolton J, Arthur D, Scroggins T, Vicini F, McCormick B, White J. RTOG 95-17, a Phase II trial to evaluate brachytherapy as the sole method of radiation therapy for Stage I and II breast carcinoma--year-5 toxicity and cosmesis. Brachytherapy. 2014 Jan-Feb;13(1):17-22. doi: 10.1016/j.brachy.2013.08.002. Epub 2013 Sep 14. PMID 24041956
- [Background] Coles CE, Griffin CL, Kirby AM, Titley J, Agrawal RK, Alhasso A, Bhattacharya IS, Brunt AM, Ciurlionis L, Chan C, Donovan EM, Emson MA, Harnett AN, Haviland JS, Hopwood P, Jefford ML, Kaggwa R, Sawyer EJ, Syndikus I, Tsang YM, Wheatley DA, Wilcox M, Yarnold JR, Bliss JM; IMPORT Trialists. Partial-breast radiotherapy after breast conservation surgery for patients with early breast cancer (UK IMPORT LOW trial): 5-year results from a multicentre, randomised, controlled, phase 3, non-inferiority trial. Lancet. 2017 Sep 9;390(10099):1048-1060. doi: 10.1016/S0140-6736(17)31145-5. Epub 2017 Aug 2. PMID 28779963
- [Background] Veronesi U, Orecchia R, Maisonneuve P, Viale G, Rotmensz N, Sangalli C, Luini A, Veronesi P, Galimberti V, Zurrida S, Leonardi MC, Lazzari R, Cattani F, Gentilini O, Intra M, Caldarella P, Ballardini B. Intraoperative radiotherapy versus external radiotherapy for early breast cancer (ELIOT): a randomised controlled equivalence trial. Lancet Oncol. 2013 Dec;14(13):1269-77. doi: 10.1016/S1470-2045(13)70497-2. Epub 2013 Nov 11. PMID 24225155
- [Background] Vaidya JS, Wenz F, Bulsara M, Tobias JS, Joseph DJ, Keshtgar M, Flyger HL, Massarut S, Alvarado M, Saunders C, Eiermann W, Metaxas M, Sperk E, Sutterlin M, Brown D, Esserman L, Roncadin M, Thompson A, Dewar JA, Holtveg HM, Pigorsch S, Falzon M, Harris E, Matthews A, Brew-Graves C, Potyka I, Corica T, Williams NR, Baum M; TARGIT trialists' group. Risk-adapted targeted intraoperative radiotherapy versus whole-breast radiotherapy for breast cancer: 5-year results for local control and overall survival from the TARGIT-A randomised trial. Lancet. 2014 Feb 15;383(9917):603-13. doi: 10.1016/S0140-6736(13)61950-9. Epub 2013 Nov 11. PMID 24224997